CLINICAL TRIAL: NCT02082626
Title: A Phase I Study of Eribulin, a Novel Microtubule Inhibitor, in Children With Refractory or Recurrent Solid Tumors
Brief Title: Study of Eribulin in Children With Cancer to Determine Safety
Acronym: ERIBULIN
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Competing study opened
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3812
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Pediatric Cancer; Solid Tumors; Lymphoma
Keywords: Phase I; Pediatric; Cancer; Lymphoma; Eribulin
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eribulin (Experimental): All patients will receive the experimental agent eribulin. The dose will increase with subsequent cohorts of patients.
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate
  Other Names: Halaven

SUMMARY:
This is a study for children with cancer with no curative treatment options. The investigators will be giving eribulin, a new chemotherapy agent, for the first time to children. This study is designed to determine a safe dose the investigators can give to children in larger studies. The investigators will be monitoring the children on this study for the safety of the treatment and levels of eribulin in the blood after treatment. The investigators will also study the effect of the agent on the cancer.

DETAILED DESCRIPTION:
This is a phase I study of eribulin, a novel tubulin inhibitor in children with relapsed and refractory solid tumors including lymphoma. Dose escalation will be performed in a classic 3+3 design starting with 75% of the adult maximum tolerated dose (MTD). Pharmacokinetics will be done on each patient. Primary endpoint will be the pediatric MTD.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 21 years of age at the time of study enrollment
* Diagnosis: refractory or recurrent solid tumors, including lymphomas, except those with CNS tumors or known CNS metastases
* Disease Status: measurable or evaluable disease
* Adequate organ function as defined in protocol

Exclusion Criteria:

* Pregnant or breastfeeding

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  The dose that does not cause dose limiting toxicity during the first cycle in more than 1 of 6 subjects

SECONDARY OUTCOMES:
Pharmacokinetics of eribulin in children with cancer | 8 days after first dose
  13 blood samples will be drawn from each subject over first 8 days of protocol to measure serum levels of the agent eribulin.
Tumor expression of BRCP and ABCB1 | 1 year
  Archival tumor samples from each subject will be stained for expression of BRCP and ABCB1, transporter proteins responsible for some resistance to chemotherapy. Will compare expression and response data
Tumor response | 2 years
  Subjects receiving eribulin will have scans approximately every 6 weeks to assess whether the tumors are growing, shrinking, or remaining stable.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Y McNall-Knapp, MD, Principal Investigator — University of Oklahoma; Amanda Linz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Jimmy Everest Center for Cancer and Blood Disorders in Children, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No